CLINICAL TRIAL: NCT00659607
Title: PMS Study of MicardisPlus Tablet
Brief Title: Telmisartan+HCTZ (Hydrochlorothiazide), Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 502.475
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Results first posted 2009-10-22 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This Post Marketing Surveillance (PMS) study aims to review the followings by investigating the actual practice of MicardisPlus Tablet on the market:

1. Unexpected adverse drug reactions (especially, serious adverse events (SAEs))
2. Frequency of incidence and its change in adverse events (AEs)
3. Factors on the safety profile of the study drug
4. Factors on the efficacy profile of the study drug

ELIGIBILITY:
Inclusion Criteria:

patients diagnosed with essential hypertension

Exclusion Criteria:

patients who took Micardis Plus before participating in this PMS study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals and clinics in Korea
Sampling Method: Probability Sample
Enrollment: 6901 (Actual)
Dates: Start 2003-09; Primary Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (326):
- South Korea (326):
  - Boehringer Ingelheim Investigational Site 10, Busan
  - Boehringer Ingelheim Investigational Site 11, Busan
  - Boehringer Ingelheim Investigational Site 12, Busan
  - Boehringer Ingelheim Investigational Site 13, Busan
  - Boehringer Ingelheim Investigational Site 14, Busan
  - Boehringer Ingelheim Investigational Site 15, Busan
  - Boehringer Ingelheim Investigational Site 16, Busan
  - Boehringer Ingelheim Investigational Site 17, Busan
  - Boehringer Ingelheim Investigational Site 18, Busan
  - Boehringer Ingelheim Investigational Site 19, Busan
  - Boehringer Ingelheim Investigational Site 1, Busan
  - Boehringer Ingelheim Investigational Site 20, Busan
  - Boehringer Ingelheim Investigational Site 21, Busan
  - Boehringer Ingelheim Investigational Site 22, Busan
  - Boehringer Ingelheim Investigational Site 23, Busan
  - Boehringer Ingelheim Investigational Site 24, Busan
  - Boehringer Ingelheim Investigational Site 25, Busan
  - Boehringer Ingelheim Investigational Site 26, Busan
  - Boehringer Ingelheim Investigational Site 27, Busan
  - Boehringer Ingelheim Investigational Site 28, Busan
  - Boehringer Ingelheim Investigational Site 29, Busan
  - Boehringer Ingelheim Investigational Site 2, Busan
  - Boehringer Ingelheim Investigational Site 30, Busan
  - Boehringer Ingelheim Investigational Site 31, Busan
  - Boehringer Ingelheim Investigational Site 32, Busan
  - Boehringer Ingelheim Investigational Site 33, Busan
  - Boehringer Ingelheim Investigational Site 34, Busan
  - Boehringer Ingelheim Investigational Site 35, Busan
  - Boehringer Ingelheim Investigational Site 36, Busan
  - Boehringer Ingelheim Investigational Site 37, Busan
  - Boehringer Ingelheim Investigational Site 38, Busan
  - Boehringer Ingelheim Investigational Site 39, Busan
  - Boehringer Ingelheim Investigational Site 3, Busan
  - Boehringer Ingelheim Investigational Site 40, Busan
  - Boehringer Ingelheim Investigational Site 41, Busan
  - Boehringer Ingelheim Investigational Site 42, Busan
  - Boehringer Ingelheim Investigational Site 43, Busan
  - Boehringer Ingelheim Investigational Site 44, Busan
  - Boehringer Ingelheim Investigational Site 45, Busan
  - Boehringer Ingelheim Investigational Site 46, Busan
  - Boehringer Ingelheim Investigational Site 47, Busan
  - Boehringer Ingelheim Investigational Site 48, Busan
  - Boehringer Ingelheim Investigational Site 49, Busan
  - Boehringer Ingelheim Investigational Site 4, Busan
  - Boehringer Ingelheim Investigational Site 5, Busan
  - Boehringer Ingelheim Investigational Site 6, Busan
  - Boehringer Ingelheim Investigational Site 7, Busan
  - Boehringer Ingelheim Investigational Site 8, Busan
  - Boehringer Ingelheim Investigational Site 9, Busan
  - Boehringer Ingelheim Investigational Site 10, Daegu
  - Boehringer Ingelheim Investigational Site 11, Daegu
  - Boehringer Ingelheim Investigational Site 12, Daegu
  - Boehringer Ingelheim Investigational Site 13, Daegu
  - Boehringer Ingelheim Investigational Site 14, Daegu
  - Boehringer Ingelheim Investigational Site 15, Daegu
  - Boehringer Ingelheim Investigational Site 16, Daegu
  - Boehringer Ingelheim Investigational Site 17, Daegu
  - Boehringer Ingelheim Investigational Site 18, Daegu
  - Boehringer Ingelheim Investigational Site 19, Daegu
  - Boehringer Ingelheim Investigational Site 1, Daegu
  - Boehringer Ingelheim Investigational Site 20, Daegu
  - Boehringer Ingelheim Investigational Site 21, Daegu
  - Boehringer Ingelheim Investigational Site 22, Daegu
  - Boehringer Ingelheim Investigational Site 23, Daegu
  - Boehringer Ingelheim Investigational Site 24, Daegu
  - Boehringer Ingelheim Investigational Site 25, Daegu
  - Boehringer Ingelheim Investigational Site 26, Daegu
  - Boehringer Ingelheim Investigational Site 27, Daegu
  - Boehringer Ingelheim Investigational Site 2, Daegu
  - Boehringer Ingelheim Investigational Site 3, Daegu
  - Boehringer Ingelheim Investigational Site 4, Daegu
  - Boehringer Ingelheim Investigational Site 5, Daegu
  - Boehringer Ingelheim Investigational Site 6, Daegu
  - Boehringer Ingelheim Investigational Site 7, Daegu
  - Boehringer Ingelheim Investigational Site 8, Daegu
  - Boehringer Ingelheim Investigational Site 9, Daegu
  - Boehringer Ingelheim Investigational Site 10, Daejeon
  - Boehringer Ingelheim Investigational Site 11, Daejeon
  - Boehringer Ingelheim Investigational Site 12, Daejeon
  - Boehringer Ingelheim Investigational Site 13, Daejeon
  - Boehringer Ingelheim Investigational Site 14, Daejeon
  - Boehringer Ingelheim Investigational Site 15, Daejeon
  - Boehringer Ingelheim Investigational Site 16, Daejeon
  - Boehringer Ingelheim Investigational Site 17, Daejeon
  - Boehringer Ingelheim Investigational Site 18, Daejeon
  - Boehringer Ingelheim Investigational Site 19, Daejeon
  - Boehringer Ingelheim Investigational Site 1, Daejeon
  - Boehringer Ingelheim Investigational Site 20, Daejeon
  - Boehringer Ingelheim Investigational Site 21, Daejeon
  - Boehringer Ingelheim Investigational Site 22, Daejeon
  - Boehringer Ingelheim Investigational Site 23, Daejeon
  - Boehringer Ingelheim Investigational Site 24, Daejeon
  - Boehringer Ingelheim Investigational Site 25, Daejeon
  - Boehringer Ingelheim Investigational Site 26, Daejeon
  - Boehringer Ingelheim Investigational Site 27, Daejeon
  - Boehringer Ingelheim Investigational Site 28, Daejeon
  - Boehringer Ingelheim Investigational Site 29, Daejeon
  - Boehringer Ingelheim Investigational Site 2, Daejeon
  - Boehringer Ingelheim Investigational Site 30, Daejeon
  - Boehringer Ingelheim Investigational Site 31, Daejeon
  - Boehringer Ingelheim Investigational Site 3, Daejeon
  - Boehringer Ingelheim Investigational Site 4, Daejeon
  - Boehringer Ingelheim Investigational Site 5, Daejeon
  - Boehringer Ingelheim Investigational Site 6, Daejeon
  - Boehringer Ingelheim Investigational Site 7, Daejeon
  - Boehringer Ingelheim Investigational Site 8, Daejeon
  - Boehringer Ingelheim Investigational Site 9, Daejeon
  - Boehringer Ingelheim Investigational Site 10, Gangwondo
  - Boehringer Ingelheim Investigational Site 11, Gangwondo
  - Boehringer Ingelheim Investigational Site 12, Gangwondo
  - Boehringer Ingelheim Investigational Site 13, Gangwondo
  - Boehringer Ingelheim Investigational Site 1, Gangwondo
  - Boehringer Ingelheim Investigational Site 2, Gangwondo
  - Boehringer Ingelheim Investigational Site 3, Gangwondo
  - Boehringer Ingelheim Investigational Site 4, Gangwondo
  - Boehringer Ingelheim Investigational Site 5, Gangwondo
  - Boehringer Ingelheim Investigational Site 6, Gangwondo
  - Boehringer Ingelheim Investigational Site 7, Gangwondo
  - Boehringer Ingelheim Investigational Site 8, Gangwondo
  - Boehringer Ingelheim Investigational Site 9, Gangwondo
  - Boehringer Ingelheim Investigational Site 10, Gwangju
  - Boehringer Ingelheim Investigational Site 11, Gwangju
  - Boehringer Ingelheim Investigational Site 12, Gwangju
  - Boehringer Ingelheim Investigational Site 13, Gwangju
  - Boehringer Ingelheim Investigational Site 14, Gwangju
  - Boehringer Ingelheim Investigational Site 15, Gwangju
  - Boehringer Ingelheim Investigational Site 16, Gwangju
  - Boehringer Ingelheim Investigational Site 17, Gwangju
  - Boehringer Ingelheim Investigational Site 18, Gwangju
  - Boehringer Ingelheim Investigational Site 19, Gwangju
  - Boehringer Ingelheim Investigational Site 1, Gwangju
  - Boehringer Ingelheim Investigational Site 20, Gwangju
  - Boehringer Ingelheim Investigational Site 21, Gwangju
  - Boehringer Ingelheim Investigational Site 22, Gwangju
  - Boehringer Ingelheim Investigational Site 23, Gwangju
  - Boehringer Ingelheim Investigational Site 24, Gwangju
  - Boehringer Ingelheim Investigational Site 25, Gwangju
  - Boehringer Ingelheim Investigational Site 26, Gwangju
  - Boehringer Ingelheim Investigational Site 27, Gwangju
  - Boehringer Ingelheim Investigational Site 28, Gwangju
  - Boehringer Ingelheim Investigational Site 29, Gwangju
  - Boehringer Ingelheim Investigational Site 2, Gwangju
  - Boehringer Ingelheim Investigational Site 30, Gwangju
  - Boehringer Ingelheim Investigational Site 31, Gwangju
  - Boehringer Ingelheim Investigational Site 32, Gwangju
  - Boehringer Ingelheim Investigational Site 33, Gwangju
  - Boehringer Ingelheim Investigational Site 34, Gwangju
  - Boehringer Ingelheim Investigational Site 35, Gwangju
  - Boehringer Ingelheim Investigational Site 36, Gwangju
  - Boehringer Ingelheim Investigational Site 37, Gwangju
  - Boehringer Ingelheim Investigational Site 38, Gwangju
  - Boehringer Ingelheim Investigational Site 39, Gwangju
  - Boehringer Ingelheim Investigational Site 3, Gwangju
  - Boehringer Ingelheim Investigational Site 40, Gwangju
  - Boehringer Ingelheim Investigational Site 41, Gwangju
  - Boehringer Ingelheim Investigational Site 42, Gwangju
  - Boehringer Ingelheim Investigational Site 43, Gwangju
  - Boehringer Ingelheim Investigational Site 4, Gwangju
  - Boehringer Ingelheim Investigational Site 5, Gwangju
  - Boehringer Ingelheim Investigational Site 6, Gwangju
  - Boehringer Ingelheim Investigational Site 7, Gwangju
  - Boehringer Ingelheim Investigational Site 8, Gwangju
  - Boehringer Ingelheim Investigational Site 9, Gwangju
  - Boehringer Ingelheim Investigational Site, Gyeongbuk
  - Boehringer Ingelheim Investigational Site 10, Gyeonggido
  - Boehringer Ingelheim Investigational Site 11, Gyeonggido
  - Boehringer Ingelheim Investigational Site 12, Gyeonggido
  - Boehringer Ingelheim Investigational Site 13, Gyeonggido
  - Boehringer Ingelheim Investigational Site 14, Gyeonggido
  - Boehringer Ingelheim Investigational Site 15, Gyeonggido
  - Boehringer Ingelheim Investigational Site 16, Gyeonggido
  - Boehringer Ingelheim Investigational Site 17, Gyeonggido
  - Boehringer Ingelheim Investigational Site 18, Gyeonggido
  - Boehringer Ingelheim Investigational Site 19, Gyeonggido
  - Boehringer Ingelheim Investigational Site 1, Gyeonggido
  - Boehringer Ingelheim Investigational Site 20, Gyeonggido
  - Boehringer Ingelheim Investigational Site 21, Gyeonggido
  - Boehringer Ingelheim Investigational Site 22, Gyeonggido
  - Boehringer Ingelheim Investigational Site 23, Gyeonggido
  - Boehringer Ingelheim Investigational Site 24, Gyeonggido
  - Boehringer Ingelheim Investigational Site 25, Gyeonggido
  - Boehringer Ingelheim Investigational Site 26, Gyeonggido
  - Boehringer Ingelheim Investigational Site 27, Gyeonggido
  - Boehringer Ingelheim Investigational Site 28, Gyeonggido
  - Boehringer Ingelheim Investigational Site 29, Gyeonggido
  - Boehringer Ingelheim Investigational Site 2, Gyeonggido
  - Boehringer Ingelheim Investigational Site 30, Gyeonggido
  - Boehringer Ingelheim Investigational Site 31, Gyeonggido
  - Boehringer Ingelheim Investigational Site 32, Gyeonggido
  - Boehringer Ingelheim Investigational Site 33, Gyeonggido
  - Boehringer Ingelheim Investigational Site 34, Gyeonggido
  - Boehringer Ingelheim Investigational Site 35, Gyeonggido
  - Boehringer Ingelheim Investigational Site 36, Gyeonggido
  - Boehringer Ingelheim Investigational Site 37, Gyeonggido
  - Boehringer Ingelheim Investigational Site 38, Gyeonggido
  - Boehringer Ingelheim Investigational Site 39, Gyeonggido
  - Boehringer Ingelheim Investigational Site 3, Gyeonggido
  - Boehringer Ingelheim Investigational Site 40, Gyeonggido
  - Boehringer Ingelheim Investigational Site 41, Gyeonggido
  - Boehringer Ingelheim Investigational Site 42, Gyeonggido
  - Boehringer Ingelheim Investigational Site 43, Gyeonggido
  - Boehringer Ingelheim Investigational Site 44, Gyeonggido
  - Boehringer Ingelheim Investigational Site 45, Gyeonggido
  - Boehringer Ingelheim Investigational Site 46, Gyeonggido
  - Boehringer Ingelheim Investigational Site 47, Gyeonggido
  - Boehringer Ingelheim Investigational Site 48, Gyeonggido
  - Boehringer Ingelheim Investigational Site 49, Gyeonggido
  - Boehringer Ingelheim Investigational Site 4, Gyeonggido
  - Boehringer Ingelheim Investigational Site 50, Gyeonggido
  - Boehringer Ingelheim Investigational Site 51, Gyeonggido
  - Boehringer Ingelheim Investigational Site 52, Gyeonggido
  - Boehringer Ingelheim Investigational Site 53, Gyeonggido
  - Boehringer Ingelheim Investigational Site 54, Gyeonggido
  - Boehringer Ingelheim Investigational Site 55, Gyeonggido
  - Boehringer Ingelheim Investigational Site 56, Gyeonggido
  - Boehringer Ingelheim Investigational Site 57, Gyeonggido
  - Boehringer Ingelheim Investigational Site 58, Gyeonggido
  - Boehringer Ingelheim Investigational Site 59, Gyeonggido
  - Boehringer Ingelheim Investigational Site 5, Gyeonggido
  - Boehringer Ingelheim Investigational Site 60, Gyeonggido
  - Boehringer Ingelheim Investigational Site 61, Gyeonggido
  - Boehringer Ingelheim Investigational Site 62, Gyeonggido
  - Boehringer Ingelheim Investigational Site 63, Gyeonggido
  - Boehringer Ingelheim Investigational Site 64, Gyeonggido
  - Boehringer Ingelheim Investigational Site 65, Gyeonggido
  - Boehringer Ingelheim Investigational Site 66, Gyeonggido
  - Boehringer Ingelheim Investigational Site 67, Gyeonggido
  - Boehringer Ingelheim Investigational Site 68, Gyeonggido
  - Boehringer Ingelheim Investigational Site 69, Gyeonggido
  - Boehringer Ingelheim Investigational Site 6, Gyeonggido
  - Boehringer Ingelheim Investigational Site 70, Gyeonggido
  - Boehringer Ingelheim Investigational Site 71, Gyeonggido
  - Boehringer Ingelheim Investigational Site 7, Gyeonggido
  - Boehringer Ingelheim Investigational Site 8, Gyeonggido
  - Boehringer Ingelheim Investigational Site 9, Gyeonggido
  - Boehringer Ingelheim Investigational Site, Gyeongnam
  - Boehringer Ingelheim Investigational Site 1, Incheon
  - Boehringer Ingelheim Investigational Site 2, Incheon
  - Boehringer Ingelheim Investigational Site 3, Incheon
  - Boehringer Ingelheim Investigational Site 4, Incheon
  - Boehringer Ingelheim Investigational Site 5, Incheon
  - Boehringer Ingelheim Investigational Site 6, Incheon
  - Boehringer Ingelheim Investigational Site 7, Incheon
  - Boehringer Ingelheim Investigational Site 8, Incheon
  - Boehringer Ingelheim Investigational Site 9, Incheon
  - Boehringer Ingelheim Investigational Site 1, Jeju City
  - Boehringer Ingelheim Investigational Site 2, Jeju City
  - Boehringer Ingelheim Investigational Site, Jeonbuk
  - Boehringer Ingelheim Investigational Site 1, Jeonnam
  - Boehringer Ingelheim Investigational Site 2, Jeonnam
  - Boehringer Ingelheim Investigational Site 3, Jeonnam
  - Boehringer Ingelheim Investigational Site 1, Jungnam
  - Boehringer Ingelheim Investigational Site 2, Jungnam
  - Boehringer Ingelheim Investigational Site 10, Seoul
  - Boehringer Ingelheim Investigational Site 11, Seoul
  - Boehringer Ingelheim Investigational Site 12, Seoul
  - Boehringer Ingelheim Investigational Site 13, Seoul
  - Boehringer Ingelheim Investigational Site 14, Seoul
  - Boehringer Ingelheim Investigational Site 15, Seoul
  - Boehringer Ingelheim Investigational Site 16, Seoul
  - Boehringer Ingelheim Investigational Site 17, Seoul
  - Boehringer Ingelheim Investigational Site 18, Seoul
  - Boehringer Ingelheim Investigational Site 19, Seoul
  - Boehringer Ingelheim Investigational Site 1, Seoul
  - Boehringer Ingelheim Investigational Site 20, Seoul
  - Boehringer Ingelheim Investigational Site 21, Seoul
  - Boehringer Ingelheim Investigational Site 22, Seoul
  - Boehringer Ingelheim Investigational Site 23, Seoul
  - Boehringer Ingelheim Investigational Site 24, Seoul
  - Boehringer Ingelheim Investigational Site 25, Seoul
  - Boehringer Ingelheim Investigational Site 26, Seoul
  - Boehringer Ingelheim Investigational Site 27, Seoul
  - Boehringer Ingelheim Investigational Site 28, Seoul
  - Boehringer Ingelheim Investigational Site 29, Seoul
  - Boehringer Ingelheim Investigational Site 2, Seoul
  - Boehringer Ingelheim Investigational Site 30, Seoul
  - Boehringer Ingelheim Investigational Site 31, Seoul
  - Boehringer Ingelheim Investigational Site 32, Seoul
  - Boehringer Ingelheim Investigational Site 33, Seoul
  - Boehringer Ingelheim Investigational Site 34, Seoul
  - Boehringer Ingelheim Investigational Site 35, Seoul
  - Boehringer Ingelheim Investigational Site 36, Seoul
  - Boehringer Ingelheim Investigational Site 37, Seoul
  - Boehringer Ingelheim Investigational Site 38, Seoul
  - Boehringer Ingelheim Investigational Site 39, Seoul
  - Boehringer Ingelheim Investigational Site 3, Seoul
  - Boehringer Ingelheim Investigational Site 40, Seoul
  - Boehringer Ingelheim Investigational Site 41, Seoul
  - Boehringer Ingelheim Investigational Site 42, Seoul
  - Boehringer Ingelheim Investigational Site 43, Seoul
  - Boehringer Ingelheim Investigational Site 44, Seoul
  - Boehringer Ingelheim Investigational Site 45, Seoul
  - Boehringer Ingelheim Investigational Site 46, Seoul
  - Boehringer Ingelheim Investigational Site 47, Seoul
  - Boehringer Ingelheim Investigational Site 48, Seoul
  - Boehringer Ingelheim Investigational Site 49, Seoul
  - Boehringer Ingelheim Investigational Site 4, Seoul
  - Boehringer Ingelheim Investigational Site 50, Seoul
  - Boehringer Ingelheim Investigational Site 51, Seoul
  - Boehringer Ingelheim Investigational Site 52, Seoul
  - Boehringer Ingelheim Investigational Site 53, Seoul
  - Boehringer Ingelheim Investigational Site 54, Seoul
  - Boehringer Ingelheim Investigational Site 55, Seoul
  - Boehringer Ingelheim Investigational Site 56, Seoul
  - Boehringer Ingelheim Investigational Site 57, Seoul
  - Boehringer Ingelheim Investigational Site 58, Seoul
  - Boehringer Ingelheim Investigational Site 59, Seoul
  - Boehringer Ingelheim Investigational Site 5, Seoul
  - Boehringer Ingelheim Investigational Site 60, Seoul
  - Boehringer Ingelheim Investigational Site 61, Seoul
  - Boehringer Ingelheim Investigational Site 62, Seoul
  - Boehringer Ingelheim Investigational Site 63, Seoul
  - Boehringer Ingelheim Investigational Site 64, Seoul
  - Boehringer Ingelheim Investigational Site 65, Seoul
  - Boehringer Ingelheim Investigational Site 66, Seoul
  - Boehringer Ingelheim Investigational Site 67, Seoul
  - Boehringer Ingelheim Investigational Site 68, Seoul
  - Boehringer Ingelheim Investigational Site 69, Seoul
  - Boehringer Ingelheim Investigational Site 6, Seoul
  - Boehringer Ingelheim Investigational Site 70, Seoul
  - Boehringer Ingelheim Investigational Site 71, Seoul
  - Boehringer Ingelheim Investigational Site 72, Seoul
  - Boehringer Ingelheim Investigational Site 73, Seoul
  - Boehringer Ingelheim Investigational Site 7, Seoul
  - Boehringer Ingelheim Investigational Site 8, Seoul
  - Boehringer Ingelheim Investigational Site 9, Seoul

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 6,901 Case Report Forms were retrieved from 281 study centers. Three thousand and nine hundred thirty two (3,932) patients were eligible for the safety assessment. As requested by KFDA to be in line with the registered indication, 2, 969 patients with mild hypertension and treatment naïve patients were excluded from analysis.
Groups:
- Hypertensive Patients With Micardis Plus for the First Time: In Post Marketing Surveillance (PMS), there are totally three figures. The number of enrolled patients: 6,901/ The number of patients for safety assessment: 3,932/ The number of patients for efficacy assessment: 3,616.
Period: Overall Study
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Started | 3932
Completed | 3616
Not Completed | 316
Not completed — No blood pressure recorded | 147
Not completed — Unknown measuring date of blood pressure | 85
Not completed — 'Unable to evaluate' for the final asses | 67
Not completed — No recorded efficacy data | 15
Not completed — Inconsistent BP measuring date | 2

BASELINE CHARACTERISTICS:
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3917
Age, Continuous [Mean (Standard Deviation); unit: years] — Date of birth not recorded for 15 patients,
  years | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender not recorded for 15 patients
  Participants
    Female | 2057
    Male | 1860

OUTCOME MEASURES:

1. Primary Outcome: Unexpected Adverse Events
Description: Occurrence status of unexpected adverse events
Time Frame: Up to 6 years
Population: Out of 6,901 patients, 3,932 patients were analyzed for the safety assessment
Measure: Number; unit: Percentage of patients
Groups:
- Hypertensive Patients With Micardis Plus for the First Time: In Post Marketing Surveillance (PMS), there are totally three figures. The number of enrolled patients: 6,901. The number of patients for safety assessment: 3932
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3932
Percentage of patients | 0.58

2. Primary Outcome: Frequency of Adverse Events
Time Frame: Up to 6 years
Population: Out of 6,901 patients, 3,932 patients were analyzed for the safety assessment
Measure: Number; unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3932
Percentage of patients | 1.04

3. Primary Outcome: Change From Baseline in SBP (Systolic Blood Pressure) at Week 2
Description: Effect on decrease in systolic blood pressure
Time Frame: Baseline and End of Study
Population: Out of 6,901 patients, 3,616 patients for the efficacy assessment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3614
mmHg | -29 (16)
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p < 0.0001, t-test for paired observations

4. Secondary Outcome: Gender Factors Affecting the Safety Profile
Description: Occurrence status of adverse events by Gender category of patients
Time Frame: Up to 6 years
Population: Out of 6,901 patients, 3,932 patients were analyzed for the safety assessment and Gender not recorded for 15 patients
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3917
Percentage of patients
  Male | 1.24 [0.79 to 1.85]
  Female | 0.88 [0.52 to 1.38]
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.2669, Chi-squared

5. Secondary Outcome: Age Factors Affecting the Safety Profile
Description: Occurrence status of adverse events by Age category of patients
Time Frame: Up to 6 years
Population: Out of 6,901 patients, 3,932 patients were analyzed for the safety assessment and Date of birth not recorded for 15 patients
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3917
Percentage of patients
  20 ≤ age < 30 | 0 [NA to NA] — Percentage of Patients with this category is 0
  30 ≤ age < 40 | 1.32 [0.16 to 4.70]
  40 ≤ age < 50 | 1.20 [0.52 to 2.34]
  50 ≤ age < 60 | 1.13 [0.58 to 1.96]
  60 ≤ age < 70 | 0.88 [0.42 to 1.62]
  ≥ 70 | 1.04 [0.48 to 1.96]
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.9674, Chi-squared

6. Secondary Outcome: Proportion of Geriatric Population Factor Affecting the Safety Profile
Description: Occurrence status of adverse events by Proportion of geriatric population of patients
Time Frame: Up to 6 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3917
Percentage of patients
  < 65 | 1.03 [0.68 to 1.51]
  >= 65 | 1.07 [0.60 to 1.76]
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.9207, Chi-squared

7. Secondary Outcome: Treatment Type Factors Affecting the Safety Profile
Description: Occurrence status of adverse events by Treatment type of patients
Time Frame: Up to 6 years
Population: Out of 6,901 patients, 3,932 patients were analyzed for the safety assessment and Treatment type not recorded for 294 patients
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3638
Percentage of patients
  In-patient | 0 [NA to NA] — Percentage of Patients with this category is 0
  Out-patient | 1.10 [0.78 to 1.51]
  In-patient and outpatient alternatively | 1.40 [0.17 to 4.96]
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.8249, Fisher Exact

8. Primary Outcome: Change From Baseline in DBP (Diastolic Blood Pressure) at Week 2
Description: Effect on decrease in diastolic blood pressure
Time Frame: Baseline and End of Study
Population: Out of 6,901 patients, 3,616 patients for the efficacy assessment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3614
mmHg | -15 (11)
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p < 0.0001, t-test for paired observations

9. Primary Outcome: Effective Rate
Description: Efficacy assessment (effective or not effective) based on a clinical judgement (1=Cured, 2=Improved, 3=Failed) as follows:
  Ⅰ. Effective (if the clinical judgement of investigator is 1 or 2=cured or improved)
  Ⅱ. Not effective (if the clinical judgement of investigator is 3=failed)
Time Frame: Baseline and End of Study
Population: Out of 6,901 patients, 3,616 patients for the efficacy assessment
Measure: Number; unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3616
Percentage of patients | 99

10. Secondary Outcome: Medical History Factors Affecting the Safety Profile
Description: Occurrence status of adverse events by medical history of patients
Time Frame: Up to 6 years
Population: Out of 6,901 patients, 3,932 patients were analyzed for the safety assessment
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3932
Percentage of patients
  With Medical history | 1.97 [1.24 to 2.96]
  Without Medical history | 0.68 [0.41 to 1.05]
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.0003, Chi-squared; Odds Ratio (OR) = 2.2, 95% CI 2-sided [1.121 to 4.151] — The estimation of Odds Ratio and 95% Confidence Interval based on the logistic regression analysis

11. Secondary Outcome: Concomitant Disease Factors Affecting the Safety Profile
Description: Occurrence status of adverse events by Concomitant disease of patients
Time Frame: Up to 6 years
Population: Out of 6,901 patients, 3,932 patients were analyzed for the safety assessment
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3932
Percentage of patients
  With Concomitant disease | 2.30 [1.49 to 3.38]
  Without Concomitant disease | 0.56 [0.32 to 0.91]
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p < 0.0001, Chi-squared; Odds Ratio (OR) = 3.3, 95% CI 2-sided [1.642 to 6.776] — The Estimation of Odds Ratio and 95% Confidence Interval based the logistic regression analysis

12. Secondary Outcome: Medical History Factors Affecting the Efficacy Profile
Description: Efficacy rate by medical characteristic of patients
Time Frame: Baseline and End of Study
Population: Out of 6,901 patients, 3,616 patients for the efficacy assessment
Measure: Number; unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3616
Percentage of patients
  With Medical history | 98.1
  Without Medical history | 99.2
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.0075, Chi-squared

13. Secondary Outcome: Previous Medication Factors Affecting the Efficacy Profile
Description: Efficacy rate by medical characteristic of patients
Time Frame: Baseline and End of Study
Population: Out of 6,901 patients, 3,616 patients for the efficacy assessment
Measure: Number; unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3616
Percentage of patients
  With Previous medication | 98.3
  Without Previous medication | 99.6
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.0007, Chi-squared

14. Secondary Outcome: Baseline Severity of Hypertension Factors Affecting the Efficacy Profile
Description: Efficacy rate by medical characteristic of patients
  Stage 1 (SBP 140~159 mmHg or DBP 90~99 mmHg) Stage 2 (SBP 160~179 mmHg or DBP 100~109 mmHg) Stage 3 (SBP ≥ 180 mmHg or DBP ≥ 110 mmHg)
Time Frame: Baseline and End of Study
Population: Out of 6,901 patients, 3,616 patients for the efficacy assessment
Measure: Number; unit: Percentage of patients
Groups:
- Hypertensive Patients With Micardis Plus for the First Time: In Post Marketing Surveillance (PMS), there are totally three figures. The number of enrolled patients: 6,901/ The number of patients for safety assessment: 3932/ The number of patients for efficacy assessment: 3616.
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3616
Percentage of patients
  Stage 1 | 98.3
  Stage 2 | 99.2
  Stage 3 | 98.3
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.0393, Chi-squared

15. Secondary Outcome: Daily Dose of Micardis® Plus Factors Affecting the Efficacy Profile
Description: Efficacy rate by medical characteristic of patients
  40/12.5mg < daily dose < 80/12.5mg - Because some physicians changed the daily dose based on patient's BP control result, this range exists
Time Frame: Baseline and End of Study
Population: Out of 6,901 patients, 3,616 patients for the efficacy assessment and Daily dose not recorded for 26 patients
Measure: Number; unit: Percentage of patients
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Number analyzed (Participants) | 3590
Percentage of patients
  40/12.5mg | 98.8
  40/12.5mg < daily dose < 80/12.5mg | 95.8
  80/12.5mg | 99.4
Statistical Analysis 1: Comparison: Hypertensive Patients With Micardis Plus for the First Time; Test type: Superiority or Other; p = 0.0245, Chi-squared

ADVERSE EVENTS:
Time Frame: Over a period of 6 years
Description: The number of patients for safety assessment is 3932.
Arm/Group | Hypertensive Patients With Micardis Plus for the First Time
Serious Adverse Events (participants affected / at risk) | 1/3932
Other Adverse Events (participants affected / at risk) | 0/3932
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hypertensive Patients With Micardis Plus for the First Time (N=3932)
Stroke (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.